CLINICAL TRIAL: NCT01414049
Title: PATency assessmENt of Grafts by Computerized tomographY in CORONARY Patients: the PATENCY-CORONARY Trial
Brief Title: Patency-Coronary Trial
Acronym: PATENCY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CE10.151
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Complications Due to Coronary Artery Bypass Graft; Graft Failure
Keywords: CABG; Off-pump CABG; Beating heart; Graft patency; Computed tomography angiography; Angiographic evaluation of coronary graft patency
MeSH Terms: interventions — Coronary Artery Bypass, Off-Pump

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- On-pump CABG (Experimental)
  Interventions: Procedure: On-pump CABG
- Off-pump CABG (Experimental)
  Interventions: Procedure: Off-pump CABG

INTERVENTIONS:
Procedure: On-pump CABG — Use of cardiopulmonary bypass (CPB) with cardioplegic arrest: on-pump CABG.
  Arms: On-pump CABG
Procedure: Off-pump CABG — CABG performed without the use of cardiopulmonary bypass (CPB) with cardioplegic arrest, surgery performed with the beating heart.
  Other Names: Beating heart
  Arms: Off-pump CABG

SUMMARY:
Heart bypass surgery is used to increase blood flow to the heart. This surgery is usually done using a heart-lung machine (on-pump surgery) allowing the surgeon to perform the procedure on a still heart. However, this heart-lung machine causes an inflammatory response and is linked with complications such as heart injury, stroke, brain injury, kidney failure, need for blood transfusions, irregular heart rhythms and death. An effective way of counteracting the effects of the heart-lung machine is to not use the pump itself, thus performing the bypass surgery with a beating heart (off-pump surgery). However, off-pump surgery is technically more difficult, possibly associated with a decrease in graft patency. The ongoing Coronary Artery Bypass Graft Off or On Pump Revascularization Study (CORONARY), is a prospective randomized clinical trial comparing bypass surgery done with and without the pump. Worldwide, 4700 patients will be included and followed up for 5 years. The proposed research project, The Patency AssessmenT of grafts pErformed iN CORONARY (PATENCY-CORONARY), is a prospective clinical trial for the evaluation of patency (or "openness") of the bypass grafts that will enrol 1200 consecutive CORONARY patients reaching their one year follow-up. Patients will undergo a non-invasive scan using X-rays to safely and quickly evaluate graft patency. The PATENCY-CORONARY trial will determine if off-pump surgery is associated with decreased graft patency at 1-year post-surgery compared to on-pump surgery when performed by skilled surgeons in different clinical settings, whether decreased graft patency is associated with adverse short and long-term outcomes, and explore other risk factors associated with decreased graft patency.

DETAILED DESCRIPTION:
Background: As Coronary Artery Bypass Grafting (CABG) aims to restore adequate blood supply to the ischemic heart, the success of the operation should depend mainly on the patency of the bypass grafts. Graft failure has consequences similar to those of native coronary artery disease: recurrent angina, myocardial infarct (MI), additional revascularization procedures, and premature death. CABG is generally performed using cardiopulmonary bypass (CPB) with cardioplegic arrest allowing the surgeon to complete the delicate coronary anastomoses on a still heart in a bloodless field. Off-pump CABG surgery using specially designed heart stabilizer systems has been proposed as a less invasive approach to CABG avoiding the CPB circuit itself. The benefits of off-pump CABG compared with conventional on-pump CABG are still intensively debated. Multislice spiral computed tomography angiography (CTA) represents a non-invasive method as compared to conventional coronary angiography allowing a comprehensive and objective imaging of bypass grafts and native coronaries with elevated diagnostic accuracy.

Rationale: CORONARY trial (NCT00463294) is a large, international, prospective, CIHR-funded, randomized controlled trial assessing both the short and long-term clinical outcomes of 4,700 patients undergoing on-pump or off-pump CABG. However, angiographic evaluation of coronary graft patency was not intended in CORONARY.

Objectives: PATENCY-CORONARY is a new prospective trial of a consecutive subset of 1,200 CORONARY patients reaching their one-year follow-up who will undergo graft patency assessment using CTA and 3D reconstructions. This trial will determine whether off-pump compared to on-pump CABG surgery is associated with lower CABG patency when performed by experienced surgeons and if there is an association between graft failure assessed by CTA, and the occurrence of CORONARY primary outcomes (composite of death, angina, MI, stroke, renal failure and new coronary revascularization [CABG or PCI]).

Primary outcome: CABG patency index (i.e. the percentage of patent [non-occluded] distal anastomoses out of the total number of distal anastomoses for all patients) at 1 year after CABG surgery by experienced surgeons; Secondary outcomes: 1) graft lesion severity on a 3-point scale at 1 year (mimicking the FitzGibbon grading ABO); and 2) percentage of patients with at least one occluded bypass graft at 1 year; Tertiary outcome: correlation between CTA findings (compromised grafts) with CORONARY primary outcomes(composite of death, angina, MI, stroke, renal failure and new coronary revascularization [CABG or PCI]), at one and five-year of follow-up post-CABG.

Methods: All CORONARY patients reaching their one-year follow-up will be included consecutively in the PATENCY-CORONARY trial until the target of 1,200 CTA is reached and reasons for exclusion will be noted prospectively to prevent selection bias. Amount of contrast agent used, radiation dose and potential morbidities during this imaging procedure will be recorded. Each CTA examination will be assessed by two experienced and blinded radiologists and each graft will be classified according to conduit type and portions: body of the graft, anastomoses and the distal native coronary bed. In addition of PATENCY-CORONARY outcome analyses, patients undergoing CTA will be compared to excluded patients (no CTA) and the overall cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

•All CORONARY (NCT00463294) patients reaching their one-year follow-up (9-24 months) will be included consecutively in the PATENCY-CORONARY trial.

Exclusion Criteria:

* Has a history of severe hypersensitivity to iodinated contrast agents;
* Has known or suspected for pheochromocytoma;
* Has severe renal impairment (estimated glomerular filtration rate, eGFR <35 mL/min/1.73 m2). Patients with eGFR 35-50 mL/min/1.73 m2 will be treated with hydratation and N-acetylcysteine (Mucomyst®) as per local protocol for contrast administration;
* Has rapid atrial fibrillation or any other cardiac rhythm that precludes reliable ECG triggering;
* Has severe congestive heart failure, New York Heart Association (NYHA) Class IV;
* Is a pregnant or lactating female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2011-08; Primary Completion 2015-01 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
CABG Patency index | 12 months
  CABG patency index (i.e. the percentage of patent [non-occluded] distal anastomoses out of the total number of distal anastomoses for all patients) at 1 year after CABG surgery by experienced surgeons.

SECONDARY OUTCOMES:
Graft lesion severity | 12 months
  Graft lesion severity on a 3-point scale at 1 year (mimicking the FitzGibbon grading ABO).
Patients with at least one occluded graft | 12 months
  Percentage of patients with at least one occluded bypass graft at 1 year.
Grafts compromised and clinical outcomes | 12 months and 5 years
  Correlation between CTA findings (compromised grafts) with clinical primary outcomes of CORONARY trial (Myocardial infarct, Stroke, death), at one and five-year of follow-up post-CABG.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Noiseux, MD, Principal Investigator — CRCHUM, Montreal University
Locations (3):
- Canada (3):
  - Libin Cardiovascular Institute of Alberta, Calgary, Alberta
  - Population Health Research Institute, Hamilton, Ontario
  - Centre Hospitalier University de Montreal, Montreal, Quebec

REFERENCES:
- See also: CORONARY trial — http://www.clinicaltrials.gov/ct2/show/NCT00463294?